CLINICAL TRIAL: NCT02722473
Title: NSE Ancillary Study of The Therapeutic Hypothermia After Nonshockable Cardiac Arrest Trial.
Acronym: NSE-HYPERION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NSE-HYPERION
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Arrest; Hypothermia; Critical Care
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted controlled temperature between 32.5 and 33.5°C (Active Comparator): Patients will be placed in targeted temperature control between 32.5 and 33.5°C for 24 hours and then slowly rewarmed for targeted temperature control between 36.5 and 37.5°C for 24 hours.
  Interventions: Biological: NSE dosage "hypothermia arm"
- Targeted controlled temperature between 36.5 and 37.5°C (Placebo Comparator): Patients will be placed in targeted temperature control between 36.5 and 37.5°C for 48 hours
  Interventions: Biological: NSE dosage "normothermia arm"

INTERVENTIONS:
Biological: NSE dosage "hypothermia arm" — There 3 dosage of NSE per patient included: day 1, day 2 and day 3 during targeted temperature management between 33° and 37°C.
  Arms: Targeted controlled temperature between 32.5 and 33.5°C
Biological: NSE dosage "normothermia arm" — There 3 dosage of NSE per patient included: day 1, day 2 and day 3 during targeted temperature management at 37°C.
  Arms: Targeted controlled temperature between 36.5 and 37.5°C

SUMMARY:
Cardiac arrest is at present a major cause of mortality as well as a cause of disability for the surviving victims.In Europe, every year counts as 300,000 cardiac arrests responsible for 250,000 deaths. Thus, less than 20 % of patients discharged home with impaired quality of life associated with symptoms of tiredness, stress, anxiety. The prognosis is related to the initial cardiac rhythm present during the initiation of resuscitation. Recent progress in the improvement of mortality and neurological outcome has been achieved over the last decade thanks to the systematic implementation of a period of targeted temperature control between 32 and 34 ° C in patients who benefited from the realization of at least one electrical external shock.

There are theoretical and clinical arguments to think that achieving the same way a period of targeted temperature control between 32 and 34 ° C in patients treated for cardiac arrest with a non- shockable rhythm on arrival can also benefit from this procedure. However other arguments are against this hypothesis including an increase in the risk of infection , worsening of the patient's hemodynamic status with no benefit to him. To answer this question, we conduce a randomized multicenter study testing the potential improvement of neurological outcome through this procedure targeted temperature control between 32.5 and 33.5 ° C in these patients.

NSE-Ancillary Study of HYPERION Trial will determine impact on neurospecific enolase (brain biomarker) of two temperature target for targeted temperature management (33°C or 37°C) after cardiac arrest in non-shockable rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest in nonshockable rhythm and
* Glasgow Coma Scale score ≤8. In patients receiving sedative therapy at ICU admission, the Glasgow Coma Scale score assessed by the emergency physician just before sedative therapy initiation is used.
* Patient must be randomized in a center which participate in the ancillary study.

Exclusion Criteria:

* No-flow time >10 min (time from collapse to initiation of external cardiac massage);
* Low-flow time >60 min (time from initiation of external cardiac massage to return of spontaneous circulation).
* Major hemodynamic instability (defined as a continuous epinephrine or norepinephrine infusion at a flow rate >1 μg/Kg/min)
* Time from cardiac arrest to study inclusion >300 min
* Moribund patient
* Child C cirrhosis of the liver
* Age <18 years
* Pregnant or breastfeeding woman
* Correctional facility inmate
* Previous inclusion in another randomized clinical trial on cardiac arrest with day-90 neurological outcome as the primary endpoint
* Patient without health insurance
* Decision by the patient or next of kin to refuse the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01-14 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
NSE level between day 1 and day 3 | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Lascarrou, MD, Study Chair — CHD Vendee
Locations (14):
- France (14):
  - Medical Surgical Intensive Care Unit, Annecy
  - Medical Intensive Care Unit, Clermont-Ferrand
  - Medical Intensive Care Unit, Dijon
  - Medical Surgical Intensive Care Unit, La Roche-sur-Yon
  - Medical Surgical Intensive Care Unit, Lens
  - Medical Surgical Intensive Care Unit, Limoges
  - Medical Surgical Intensive Care Unit, Montauban
  - Medical Intensive Care Unit, Nantes
  - Medical Surgical Intensive Care Unit, Orléans
  - Medical Intensive Care Unit, Poitiers
  - Medical Surgical Intensive Care Unit, Rodez
  - Medical Surgical Intensive Care Unit, Saint-Brieuc
  - Medical Surgical Intensive Care Unit, St-Malo
  - Medical Intensive Care Unit, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lascarrou JB, Miailhe AF, le Gouge A, Cariou A, Dequin PF, Reignier J, Coupez E, Quenot JP, Legriel S, Pichon N, Thevenin D, Boulain T, Frat JP, Vimeux S, Colin G, Desroys du Roure F. NSE as a predictor of death or poor neurological outcome after non-shockable cardiac arrest due to any cause: Ancillary study of HYPERION trial data. Resuscitation. 2021 Jan;158:193-200. doi: 10.1016/j.resuscitation.2020.11.035. Epub 2020 Dec 8. PMID 33301887
- See also: Trial Protocol published in SJTREM — http://sjtrem.biomedcentral.com/articles/10.1186/s13049-015-0103-5